CLINICAL TRIAL: NCT05082350
Title: Clinical Trial to Evaluate the Efficacy of Black Garlic in Reducing Cardiovascular Risk in Subjects With Hypercholesterolemia
Brief Title: Nutritional Intervention With Black Garlic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maria Pilar Zafrilla Rentero (Other)
Collaborators: Instituto de Investigación y formación agraria y pesquera (IFAPA) (Unknown)
Responsible Party: Sponsor-Investigator, Maria Pilar Zafrilla Rentero, Vicedean of Pharmacy Degree, Catholic University of Murcia
Organization: Catholic University of Murcia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CFE/IF/28-20
Record Dates: First submitted 2021-06-08; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Hypercholesterolemia; Hypertension; Hyperlipidemias; Inflammation; Endothelial Dysfunction
Keywords: black garlic; sulphur bioactive compounds; hypercholesterolemia; hyperlipemia; inflammation; endothelial dysfunction
MeSH Terms: conditions — Hypercholesterolemia; Hypertension; Hyperlipidemias; Inflammation

STUDY DESIGN:
Intervention Model Description: A controlled clinical intervention study is proposed to determine the effect of black garlic consumption on biomarkers of cardiovascular function and associated pathologies in a healthy population at risk for cardiovascular disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Group, (Experimental): Daily consumption of 4 cloves of black garlic, not cooked, during 12 weeks
  Interventions: Dietary Supplement: black garlic
- Hypercholesterolemia (Experimental): Daily consumption of 4 cloves of black garlic, not cooked, during 12 weeks
  Interventions: Dietary Supplement: black garlic

INTERVENTIONS:
Dietary Supplement: black garlic — Daily consumption of 4 cloves of black garlic, not cooked, during 12 weeks

SUMMARY:
A controlled clinical intervention study is proposed to determine the effect of black garlic consumption on biomarkers of cardiovascular function and associated pathologies in a healthy population at risk for cardiovascular disease. Black garlic is the result of a fermentation process of common white garlic in which the temperature and humidity are kept constant over a long period of time. Black garlic is particularly rich in phenolic compounds such as S-allylcysteine or S-allyl-mercaptocysteine, with antioxidant action. It also provides vitamin C and other valuable antioxidant substances such as flavonoids.

DETAILED DESCRIPTION:
A parallel, controlled clinical trial will be performed to assess the effect of garlic on mild hypercholesterolemia.

The study will conducted in two groups of volunteer: healthy and at cardiovascular risk (hypercholesterolemic subjects), consuming black garlic, with each individual acting as its own control. The study will have a total duration of 18 weeks, divided in two stages:

* Stage 1: basal or washout stage of 2 weeks, in which volunteer follow their usual diet with restrictions
* Stage 2: intervention stage of 16 weeks, in which volunteer consume black garlic Sixty healthy volunteers (men and women) between 40-65 years old and BMI between 24.9-29.9 kg/m2 will be recruited. From the total of volunteer, 30 will correspond to the Healthy Group, which should have total blood cholesterol levels less than 200 mg/dL and LDL-cholesterol less than 135 mg/dL.

The other 30 volunteers correspond to the Cardiovascular Risk Group, which should have total cholesterol levels between 200-300 mg/dL and LDL-cholesterol levels between 135-175 mg/dL.

Other inclusion criteria established for all volunteers are: no acute or chronic pathology, (except hypercholesterolemia for the risk group), no taking drugs, hormones or dietary supplements, no smoking, no pregnancy, no vegetarianism.

The study has been approved by the Ethical Committee of Catholic University of Murcia (UCAM) and will be carried out in accordance with the Helsinki Declaration of Human Studies. Recruitment will take place at various Health Centers and at UCAM. All participants will be informed on the characteristics of the study and, after signing the informed consent, a routine analysis will be requested to classify the volunteer in the healthy or cardiovascular risk group.

To avoid bias due to gender, the number of women and men recruited in both groups will be balanced. The size of the study population has been estimated taking total blood cholesterol level as the main variable and taking into account that the study design is randomized and parallel. Considering a statistical power of 80%, a statistical significance level of 5% (one tail), a standard deviation of 6.5, aiming to estimate a difference of 2.5, the number of volunteers required is 25 for each group, rising to 30 in anticipation of dropouts. This number, being two study groups, will allow obtaining results with statistical significance in other biochemical parameters that would be determined as secondary variables of the study and that would inform on the effect of black garlic consumption on cardiovascular function and associated dysfunctions (inflammation, hypertension, endothelial function, diabetes, etc.).

After an initial washout (basal) stage common to all groups, in which the volunteers will consume their usual diet with restriction in the consumption of fresh garlic and garlic products, the intervention will start, with the consumption of black garlic for 12 weeks. Volunteers will be provided with black garlic and they will ensure that no other type of garlic or culinary seasoning is used.

Dietary and physical activity questionnaire according to the "Global Physical Activity Questionnarie (GPAQ)" will be compiled in order to collect information on habits and lifestyle, as well as to ensure the compliance of food restrictions.

During the study, visits will be scheduled on the first day and last day of each stage. The subjects will come to the Unit on fasting conditions and will provide the first morning urine. Blood sample will be taken, plasma aliquoted and stored at -80°C until analysis.

ELIGIBILITY:
Inclusion Criteria:

Healthy Group:

* Total blood cholesterol levels of less than 200 mg/dL
* LDL-cholesterol levels of less than 135 mg/dL
* Not suffer from any other pathology.
* No drugs, hormones or dietary supplements, no smoking, no pregnancy, no vegetarianism, etc.

Cardiovascular Risk Group:

* Total cholesterol levels between 200-300 mg/dL
* LDL-cholesterol levels between 135-175 mg/dL.
* No acute or chronic pathology, except hypercholesterolemia
* No drugs, hormones or dietary supplements, no smoking, no pregnancy, no vegetarianism, etc.).

Exclusion Criteria:

* Failure to meet any of the inclusion criteria

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Impact on blood pressure | changes observed from baseline at day 0 compared to 12 weeks.
  Blood pressure (diastolic, systolic)
Impact on lipid profile | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of total cholesterol, HDL, LDL, VLDL (very low-density lipoprotein), triglycerides, apolipoproteins A1 and B.

SECONDARY OUTCOMES:
Impact on blood cells (Hematology) | changes observed from baseline at day 0 compared to 12 weeks.
  Blood counts
evaluation of liver function to determine product safety | changes observed from baseline at day 0 compared to 12 weeks.
  Hepatic enzymes (GOT, GPT)
Changes in cytokine levels | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of pro-inflammatory: IL-1β, IL6 , TNF-α (tumor necrosis factor) and anti-inflammatory (IL-10, IL-17) cytokines.
Changes in chemokine MCP-1 (monocyte chemotactic protein) | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of chemokine MCP-1
Changes in C reactive protein | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of C reactive protein
Impact on endothelial function | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of nitric oxide, adhesion molecules VCAM-1 (vascular endothelial cell adhesion molecule), ICAM-1 (intercellular adhesion molecule), chemokines as markers of endothelium (E-selectin) and platelet (P-selectin) activation.
Impact on glucose levels | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of glucose
Impact on glycosylated hemoglobin (HbA1c) | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of glycosylated hemoglobin
Impact in hormones related to metabolism | changes observed from baseline at day 0 compared to 12 weeks.
  Plasma levels of thyroid hormones (TSH, T3, T4).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Murcia (UCAM), Murcia, Spain

IPD SHARING:
Plan to Share IPD: No